CLINICAL TRIAL: NCT00559104
Title: High-Dose Therapy and Autologous Stem Cell Transplantation During Remission in Poor-Risk Age-Adjusted International Prognostic Index High and High-Intermediate Risk Group Patients With Intermediate Grade and High-Grade Non-Hodgkin's Lymphoma Including Mantle Cell Lymphoma
Brief Title: Combination Chemotherapy With or Without Total-Body Irradiation Followed By Stem Cell Transplant in Treating Patients With Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 97133; P30CA033572 (NIH); CHNMC-97133 (Other: City of Hope); CDR0000573523 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Results first posted 2015-08-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-07

CONDITIONS: Lymphoma
Keywords: stage III adult diffuse mixed cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV mantle cell lymphoma; stage III mantle cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma | interventions — Carmustine; Cyclophosphamide; Etoposide; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Irradiation in conditioning (Active Comparator): total-body irradiation, etoposide, cyclophosphamide, infusion of peripheral blood stem cells, granulocyte-colony stimulating factor (G-CSF), autologous hematologic stem cell transplantation, peripheral blood stem cell transplantation
  Interventions: Drug: cyclophosphamide; Drug: etoposide; Procedure: autologous hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: total-body irradiation; Drug: G-CSF
- Carmustine in conditioning (Active Comparator): Carmustine, etoposide, cyclophosphamide, infusion of peripheral blood stem cells, granulocyte-colony stimulating factor (G-CSF), autologous hematopoietic stem cell transplantation, peripheral blood stem cell transplantation
  Interventions: Drug: carmustine; Drug: cyclophosphamide; Drug: etoposide; Procedure: autologous hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Drug: G-CSF

INTERVENTIONS:
Drug: carmustine — Unique to the Carmustine in Conditioning arm
  Other Names: BCNU
  Arms: Carmustine in conditioning
Drug: cyclophosphamide — Used in Both Arms
  Other Names: Cytoxan, CTX
Drug: etoposide — Used in Both Arms
  Other Names: VP-16
Procedure: autologous hematopoietic stem cell transplantation — Both arms are given autologous stem cell transplantation
Procedure: peripheral blood stem cell transplantation — Both arms are given peripheral blood stem cell transplantation (Peripheral blood stem cells are the material, autologous transplant is the modality).
Radiation: total-body irradiation — Unique to the Radiation in Conditioning Arm
  Arms: Irradiation in conditioning
Drug: G-CSF — G-CSF is given in both treatment arms, both to mobilize stem cells before apheresis, and to promote recovery of granulocytes after stem-cell re-infusion.
  Other Names: Granulocyte-colony stimulating factor

SUMMARY:
RATIONALE: Giving chemotherapy and radiation therapy to the entire body before an autologous peripheral stem cell transplant stops the growth of cancer cells by stopping them from dividing or killing them. The patient's stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy and radiation therapy.

PURPOSE: This phase II trial is studying the side effects of giving combination chemotherapy together with or without total-body irradiation followed by a stem cell transplant and to see how well it works in treating patients with non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the outcome of patients with poor-risk, age-adjusted International Prognostic Index high- and high-intermediate-risk, intermediate- and high-grade non-Hodgkin lymphoma undergoing high-dose therapy comprising etoposide and cyclophosphamide, either carmustine or total-body irradiation, and autologous stem cell transplantation (ASCT) given as a consolidation therapy.
* To evaluate the role of high-dose therapy and ASCT during first partial or complete remission (1PR/CR) in patients with poor-risk primary mediastinal large cell lymphoma.
* To evaluate the role of high-dose therapy and ASCT during first 1PR/CR in patients with advanced-stage mantle cell lymphoma.
* To evaluate the short-term and long-term toxicities of high-dose therapy and ASCT when performed during 1PR/CR in patients with poor-risk aggressive lymphomas.

OUTLINE: Patients are stratified according to disease (diffuse mixed, diffuse large cell, and immunoblastic lymphoma vs primary mediastinal large cell lymphoma vs small noncleaved cell lymphoma vs stage IV mantle cell lymphoma).

Patients' peripheral blood stem cells (PBSC) are collected after mobilization. A minimum of 2.0 x 10^6 CD34+ cells/kg must be collected. Patients experiencing disease progression during stem cell collection will be removed from study. Patients are assigned to undergo 1 of 2 therapeutic regimens.

* Regimen 1: Patients undergo total-body irradiation (TBI) on days -8 to -5 and receive etoposide IV over 4 hours on day -4 and cyclophosphamide IV over 2 hours on day -2. Patients undergo autologous PBSC transplantation on day 0.
* Regimen 2 (for patients who have received any prior thoracic irradiation or patients who underwent previous irradiation that precludes the use of TBI): Patients receive carmustine IV over 2 hours on days -7 to -5. Patients then receive etoposide and cyclophosphamide and undergo autologous PBSC transplantation as in regimen 1.

Patients with residual bulky disease greater than 5 cm may undergo involved-field radiotherapy before or after transplantation.

Patients are followed at days 7, 14, 21, 100 and 180 after PBSC transplantation, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* DISEASE CHARACTERISTICS:
* Biopsy-proven diagnosis of high-grade (small noncleaved cell lymphoma [SNCCL] or immunoblastic lymphoma) or intermediate-grade non-Hodgkin lymphoma (NHL) including mantle cell lymphoma (MCL)
* SNCCL patients with all of the following factors at presentation of disease:

  * Lactate dehydrogenase (LDH) > 500 IU/L
  * Unresectable bulky mass > 10 cm
  * Stage IV disease with bone marrow involvement
* MCL Patients with stage IV disease or in International Prognostic Index (IPI) high- or high-intermediate-risk group at the time of diagnosis
* Considered at diagnosis to be high- (3 risk factors) or high-intermediate-risk (2 risk factors) based on an age-adjusted IPI
* Poor prognostic factors at diagnosis include stage III or IV disease, lactate dehydrogenase (LDH) level above normal, or ECOG performance status (PS) 2-4
* Patients with primary mediastinal large cell lymphoma with or without sclerosis who at diagnosis had elevated LDH level with bulky mediastinal mass > 10 cm associated with a pleural effusion on chest radiography or computer tomography, or who have persistent mediastinal mass with positive disease by post-treatment gallium GA 67 scan
* Must have attained a complete response or partial response to first-line standard conventional chemotherapy
* ECOG PS 0-1 OR Karnofsky PS 80-100%
* Serum creatinine < 1.5 mg/dL OR creatinine clearance > 60 mL/min
* FEV_1 > 65% of predicted measurement or DLCO ≥ 45% of predicted measurement
* Cardiac ejection fraction > 50% by echocardiogram
* Bilirubin ≤ 1.5 x normal
* SGOT or SGPT ≤ 2 x normal

Exclusion Criteria:

* Evidence of lymphoma or < 10% lymphomatous involvement of bone by bilateral bone marrow aspiration and biopsy
* Abnormal cytogenetic study of bone marrow aspirate sample NOTE: A new classification scheme for adult non-Hodgkin lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.
* Positive HIV antibody
* Prior malignancies except for adequately treated basal cell or squamous cell carcinoma of the skin
* Hepatitis B surface antigen positivity
* Prior bone marrow transplantation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior bone marrow transplantation

Ages: 16 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 1998-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Auayporn P. Nademanee, MD, Study Chair — City of Hope Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Good Samaritan Regional Medical Center, Phoenix, Arizona
  - City of Hope National Medical Center--Main Campus, Duarte, California

REFERENCES:
- [Background] Nademanee A, Molina A, Dagis A, Snyder DS, O'Donnell MR, Parker P, Stein A, Smith E, Planas I, Kashyap A, Spielberger R, Fung H, Krishnan A, Bhatia R, Wong KK, Somlo G, Margolin K, Chow W, Sniecinski I, Vora N, Slovak M, Niland JC, Forman SJ. Autologous stem-cell transplantation for poor-risk and relapsed intermediate- and high-grade non-Hodgkin's lymphoma. Clin Lymphoma. 2000 Jun;1(1):46-54. doi: 10.3816/clm.2000.n.004. PMID 11707813

RESULTS

PARTICIPANT FLOW:
Groups:
- TBI-based Conditioning: total-body irradiation, etoposide, cyclophosphamide, infusion of peripheral blood stem cells, granulocyte-colony stimulating factor
  cyclophosphamide
  etoposide
  autologous hematopoietic stem cell transplantation
  peripheral blood stem cell transplantation
  total-body irradiation
  G-CSF
- nonTBI-based Conditioning: Carmustine, etoposide, cyclophosphamide, infusion of peripheral blood stem cells, granulocyte-colony stimulating factor
  carmustine
  cyclophosphamide
  etoposide
  autologous hematopoietic stem cell transplantation
  peripheral blood stem cell transplantation
  G-CSF
Period: Overall Study
Arm/Group | TBI-based Conditioning | nonTBI-based Conditioning
Started | 55 | 5
Completed | 46 (Progression was the reason for off-treatment for 9 of 9 patients who went off of treatment.) | 5
Not Completed | 9 | 0
Not completed — Lack of Efficacy | 9 | 0

BASELINE CHARACTERISTICS:
Groups:
- Irradiation in Conditioning: total-body irradiation, etoposide, cyclophosphamide, infusion of peripheral blood stem cells, granulocyte-colony stimulating factor
  cyclophosphamide
  etoposide
  autologous hematopoietic stem cell transplantation
  peripheral blood stem cell transplantation
  total-body irradiation
  G-CSF
- Carmustine in Conditioning: Carmustine, etoposide, cyclophosphamide, infusion of peripheral blood stem cells, granulocyte-colony stimulating factor
  carmustine
  cyclophosphamide
  etoposide
  autologous hematopoietic stem cell transplantation
  peripheral blood stem cell transplantation
  G-CSF
- Total: Total of all reporting groups
Arm/Group | Irradiation in Conditioning | Carmustine in Conditioning | Total
Number analyzed (Participants) | 55 | 5 | 60
Age, Continuous [Median (Full Range); unit: years] | 44.2 [19.0 to 57.7] | 32.4 [21.7 to 59.6] | 42.5 [19.0 to 59.6]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 5 | 60
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 3 | 25
  Male | 33 | 2 | 35
Region of Enrollment [Number; unit: participants]
  United States | 55 | 5 | 60

OUTCOME MEASURES:

1. Primary Outcome: Progression
Description: Event will be recorded if it occurs any time post-transplant, until date of death, last recorded contact, or end-of-study; whichever comes first.
  Below is reported Progression-free Survival: event is relapse or progression, or death.
Time Frame: Assessed at date of progression post-transplant
Population: per protocol
Measure: Number; unit: participants
Arm/Group | Irradiation in Conditioning | Carmustine in Conditioning
Number analyzed (Participants) | 55 | 5
participants | 22 | 1
Statistical Analysis 1: Comparison: Irradiation in Conditioning vs Carmustine in Conditioning; There is no power calculation as this is a phase II study. This is an Event-free Survival, in which an event can be Relapse/Progression, or Death. Censoring can be at the End of follow-up date, or at the End of study date; Test type: Superiority or Other; p = 0.51, Regression, Cox; Cox Proportional Hazard = 0.51, 95% CI 2-sided [0.07 to 3.79] — Parameter Dispersion Type: Standard Error of the Parameter Estimate, not of the mean. Standard Error = 1.02475

2. Primary Outcome: Mortality
Description: Event will be recorded if it occurs any time from the date of transplant until the end-of-study date, or the date of last contact, whichever comes first.
Time Frame: Assessed at date of death post-transplant
Population: per protocol
Measure: Number; unit: participants
Arm/Group | Irradiation in Conditioning | Carmustine in Conditioning
Number analyzed (Participants) | 55 | 5
participants | 19 | 1
Statistical Analysis 1: Comparison: Irradiation in Conditioning vs Carmustine in Conditioning; Phase II analysis: There was no power calculation; Test type: Superiority or Other; p = 0.69, Regression, Cox; Cox Proportional Hazard = 0.66, 95% CI 2-sided [0.09 to 4.99] — Numerator: Carmustine in the conditioning. Denominator: Irradiation in the conditioning. Parameter: Hazard ratio. Dispersion: Standard Error of the Hazard Ratio

3. Secondary Outcome: Short-term and Long-term Treatment-related Toxicities
Description: Patient may be assessed for toxicities any time after transplant, up to death, last contact date, or end-of-study date.
Time Frame: Any time after transplant
Population: per protocol
Measure: Number; unit: participants
Arm/Group | Irradiation in Conditioning | Carmustine in Conditioning
Number analyzed (Participants) | 55 | 5
participants | 39 | 1

ADVERSE EVENTS:
Arm/Group | Irradiation in Conditioning | Carmustine in Conditioning
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/5
Other Adverse Events (participants affected / at risk) | 39/55 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irradiation in Conditioning (N=55) | Carmustine in Conditioning (N=5)
Dermatologic (Skin) (COH) (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hepatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Mucositis (Gastrointestinal disorders) | 10 (10) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (7) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Packed red blood cell transfusion (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Platelet transfusion (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 12 (12) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (7) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 4 (4) | 0 (0)
Fever (General disorders) | 3 (3) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0)
Oedema NOS (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0)
Catheter related infection (Infections and infestations) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Infection NOS (Infections and infestations) | 1 (1) | 0 (0)
Infection, Bacterial (COH) (Infections and infestations) | 2 (2) | 0 (0)
Infection, Fungal (COH) (Infections and infestations) | 1 (1) | 0 (0)
Infection, Viral (COH) (Infections and infestations) | 1 (1) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Hyperbilirubinemia (Investigations) | 1 (1) | 0 (0)
Laboratory test abnormal (Investigations) | 1 (2) | 0 (0)
Leukopenia (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 0 (0)
Blood urine present (Renal and urinary disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No